CLINICAL TRIAL: NCT02630810
Title: Early Versus Late Oral Hydration After Cesarean Section: A Randomized Controlled Study
Brief Title: Early Versus Late Hydration After Cesarean Section (CS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, AMR HELMY YEHIA, Lecturer in Obstetrics and Gynaecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EVLHACS 1
Record Dates: First submitted 2015-12-10; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Gastrointestinal Motility and Defaecation Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early oral hydration (Experimental): Early oral intake of 100 ml clear unsweetened water 1 hour following the Cesarean Section, then upon patient's desire, then starting semisolid, solid food when participant passed flatus.
  Interventions: Other: Early oral hydration
- Delayed oral hydration (Active Comparator): Oral intake of 100 ml clear unsweetened water after 6 hours from the end of CS then upon patient's request,then starting semisolid, solid food when participant passed flatus.
  Interventions: Other: Delayed oral hydration

INTERVENTIONS:
Other: Early oral hydration — starting oral hydration 1 hour following Cesarean Section using 100 ml clear water
  Arms: Early oral hydration
Other: Delayed oral hydration — starting oral hydration 6 hours following Cesarean Section using 100 ml clear water
  Arms: Delayed oral hydration

SUMMARY:
This study evaluates the effect of early oral hydration on bowel movement after CS, it includes 2 groups: study group participants receive 100 ml water after 1hr from the end of CS, while the others receive water after 6hrs from the end of CS.

DETAILED DESCRIPTION:
Traditionally, oral intake after CS was depend on insurance of intestinal movement, since uncomplicated CS does not affect the intestine and the mother needs to care of her infants, lactates, discharged from hospital, early oral hydration may enhance bowel movement, so the investigators need to evaluate the safety of early oral hydration after CS.

This study compare the effects of introducing water during the 1st hour or after 6 hours on bowel movement after CS.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated elective or emergency lower segment Caesarean section
* average blood loss during and after cs
* regional anaesthesia
* primary or recurrent CS

Exclusion Criteria:

* surgical complications esp; intestinal injury
* postpartum hemorrhage
* medical disorder with pregnancy eg. hypertension, diabetes mellitus
* factors that may increase risk of postpartum hemorrhage as twins pregnancy, polyhydramnios and anemia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to 1st audible intestinal sound | First 12 hours after Cesarean Section
  Auscultating intestinal sounds (using stethoscope) hourly for the first 12 hours after Cesarean Section till intestinal sounds are audible.

SECONDARY OUTCOMES:
Time to passage of first flatus | Up to 48 hours following the Cesarean Section
  Recording the timing of passage of first flatus following Cesarean Section (up to the first 48 hours).
Time to first bowel motion | Up to 3 days (72 hours) following Cesarean Section
  Recording the first time the pass stools after cesarean section (up to the first 72 hours).
time to 1st breast feed | First 24 hours after the Cesarean Section
  Recording the first time to breastfeed after cesarean section (up to the first 24 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Amr Yehia, Lecturer, Principal Investigator — ainshams maternity hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No